CLINICAL TRIAL: NCT06907641
Title: Comparative Performance of 64Copper [64Cu]-SAR-bis-PSMA vs 68Ga PSMA-11 PET CT for the Detection of Prostate Cancer Recurrence in the Setting of Biochemical Failure Following Radical Prostatectomy
Acronym: Co-PSMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Collaborators: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Principal Investigator, Louise Emmett, Professor, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP11 (Co-PSMA); CT-2024-CTN-06035-1 (Other: Therapeutic Goods Administration)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer (Post Prostatectomy)
Keywords: Prostate Cancer; Salvage Radiotherapy; Prostatectomy; Co-PSMA; CLP11; Prostate Cancer Recurrence; Biochemical Failure; Radical Prostatectomy; Copper; PET scan
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 64Cu-SAR-bisPSMA (Experimental): 200MBq 64Cu-SAR-bisPSMA
  Interventions: Drug: 64Cu-SAR-bisPSMA

INTERVENTIONS:
Drug: 64Cu-SAR-bisPSMA — All participants will receive a single administration of 200 MBq of 64Cu-SAR-bisPSMA

SUMMARY:
The goal of this clinical trial is to compare 64Cu-SAR-bisPSMA PET/CT and 68Ga PSMA-11 PET/CT in men with biochemical failure following radical prostatectomy. The main questions it aims to answer are:

* Is there a difference in the number of lesions of prostate cancer recurrence detected between the 64Cu-SAR-bisPSMA PET/CT and 68Ga PSMA-11 PET/CT scans.
* What is the diagnostic accuracy of 64Cu-SAR-bisPSMA PET/CT compared to 68Ga PSMA-11 PET/CT using a standard of care comparator.
* Evaluate the magnitude of clinical management change when using 64Cu-SAR-bisPSMA additional to standard of care imaging (68Ga PSMA-11).

Participants will:

* have 3 visits: 1) standard of care 68Ga PSMA-11 dose and PET/CT scan; 2) 64Cu-SAR-bisPSMA dose and PET/CT; 3) 64Cu-SAR-bisPSMA PET/CT only
* have standard of care blood test either at Visit 1 or Visit 2

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 or above
* Ability to provide informed consent documentation indicating that they understand the purpose of, and procedures required for the study, and are willing to participate in the study.
* Prior radical prostatectomy for confirmed adenocarcinoma on histopathology.
* Rising PSA (0.20 - 0.75 ng/mL) following radical prostatectomy with no prior salvage radiotherapy.
* 68Ga PSMA-11 PET/CT within the last 4 weeks for prostate cancer biochemical recurrence.

Exclusion Criteria:

* Prior, or contraindication to, salvage radiotherapy for biochemically recurrent prostate cancer.
* History of current active malignancy as per investigator discretion other than prostate cancer.
* Known or expected hypersensitivity to 64Cu-SAR-bisPSMA
* Systemic therapy for metastatic prostate cancer including androgen deprivation therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients
Enrollment: 50 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Detection rate of lesions per participants, between 64Cu-SAR-bisPSMA and 68Ga PSMA-11 PET/CT | 12 months
  Compare the detection rate of sites of prostate cancer recurrence, as determined by number of lesions per participants, between 64Cu-SAR-bisPSMA and 68Ga PSMA-11 PET/CT in patients with biochemical recurrence following radical prostatectomy who are being considered for curative salvage radiotherapy.

SECONDARY OUTCOMES:
Compare the number of lesions outside of the prostatic fossa per patient between 64Cu-SAR-bisPSMA and 68Ga PSMA-11 PET/CT. | 12 months
Compare the diagnostic accuracy of 64Cu-SAR-bisPSMA versus 68Ga PSMA-11 PET/CT in the detection of recurrent or metastatic prostate cancer using a composite standard of truth | 12 months
  Compare the diagnostic accuracy of 64Cu-SAR-bisPSMA versus 68Ga PSMA-11 PET/CT in the detection of recurrent or metastatic prostate cancer using a composite standard of truth (biopsy, concurrent imaging and response to targeted therapy).
Evaluate the magnitude of clinical management change when using 64Cu-SAR-bisPSMA additional to standard of care imaging (68Ga PSMA-11). | 12 months
Compare the total number of lesions between 1 to 4-hour, and 24-hour 64Cu-SAR-bisPSMA PET/CT imaging timepoints. | 12 months
Evaluate the frequency of prostatic fossa recurrence on the 24-hour 64Cu-SAR-bisPSMA images compared to the 1 to 4-hour 64Cu-SAR-bisPSMA and 1-hour 68Ga PSMA-11 PET/CT images | 12 months
Evaluate biochemical (PSA) response following salvage radiotherapy by 64Cu-SAR-bisPSMA and 68Ga PSMA-11 PET/CT imaging parameters in the presence of normal testosterone levels. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's Hospital, Sydney, Darlinghurst, New South Wales, Australia